CLINICAL TRIAL: NCT01462461
Title: Pilot Study of the Efficacy of a Virtual Integrated Environment in Decreasing Phantom Limb Pain
Brief Title: Virtual Integrated Environment in Decreasing Phantom Limb Pain
Acronym: VIE
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 20448; W81XWH-09-2-0148 (Other Grant/Funding Number: Henry M. Jackson Foundation)
Record Dates: First submitted 2011-10-25; First posted 2011-10-31 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Phantom Limb
Keywords: Phantom Limb; Amputation, Traumatic; Electromyography; Visual Analog Pain Scale
MeSH Terms: conditions — Phantom Limb; Amputation, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if observing a virtual arm decreases phantom limb pain (PLP) in upper extremity amputees.

DETAILED DESCRIPTION:
Nearly all traumatic limb amputees will experience cognizance of a phantom limb and perceive a vivid impression that their lost limb is not only fully present, but also painful. The John Hopkins University Applied Physics Laboratory Virtual Integration Environment (VIE) is a highly flexible and adaptable virtual reality system that allows patients to observe movement of a 3D virtual arm. Using the VIE, recorded signals from the residual limb will be correlated to the desired motion of the phantom limb. We hope to correlate the consistency of these patterns with PLP to determine if increased control of the phantom limb leads to decreased PLP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 65 years of age, active duty military, beneficiary, or retiree.
* Written informed consent and written authorization for use or release of health and research study information.
* At least one upper-limb amputation (trans radial or trans humeral) at any time prior to enrollment.
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* Normal neurological examination with the exception of limb amputation.
* Ability to follow study instructions and likely to complete all required visits.
* Experiencing PLP at least 3 times a week at an intensity of at least 3 out of 10 at the time of enrollment.

Exclusion Criteria:

* Presence of mild to severe traumatic brain injury - permanent or temporary impairments of cognitive, physical, and psychosocial functions with an associated diminished or altered state of consciousness - as indicated by neuropsychological screening that is currently performed routinely on patients by the traumatic brain injury (TBI) program at Walter Reed National Military Medical Center (WRNMMC) and noted in the patient's medical record.
* Known uncontrolled systemic disease
* Participation (either concurrently or in the 30 days prior to enrollment) in another study for treatment of PLP
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound study results, or interfere significantly with the subject's participation in the study.
* Significant Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study
* Subjects with lack of effort as determined by the neurologist or psychiatrist. Subjects will be screened for effort using the Test of Memory Malingering (TOMM) in order to exclude those with blatant exaggeration or malingering. Subjects who score lower than 42/50 on the TOMM-2 will not continue in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seven unilateral, upper-extremity amputees completed the study. These subjects were either trans-radial (n=4) or trans-humeral (n=3) amputees.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Phantom Limb Pain Severity | Baseline (0 weeks) and 4 weeks
  Severity of PLP will be assessed using the Visual Analog Scale (VAS), which wil consist of a 10-cm horizontal line across which subjects will place a mark corresponding to the level of phantom limb pain he or she experiences. The distance in centimeters from the low end of the VAS to the subject's mark will be used as a numeric index of pain severity. The VAS score over 4 weeks of VIE treatment will be averaged and compared to the baseline VAS score at the start of treatment.

SECONDARY OUTCOMES:
Consistency of sEMG recordings | Baseline (0 weeks) and 4 weeks
  The activation patterns of muscles on an around the residual limb will be recorded during the initial VIE therapy session using surface electrodes. The sEMG recordings after 4 weeks will be compared to the initial sEMG recordings at the start of VIE treatment. The change in sEMG signals over time will indicate how well patients are able to replicate muscle activation patterns between sessions in which they attempt to move the phantom arm in the same manner as the virtual arm.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Pasquina, MD, MC, Principal Investigator — Walter Reed National Military Medical Center (WRNMMC)
Locations (1):
- Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Ramachandran VS, Hirstein W. The perception of phantom limbs. The D. O. Hebb lecture. Brain. 1998 Sep;121 ( Pt 9):1603-30. doi: 10.1093/brain/121.9.1603. PMID 9762952
- [Background] Carlen PL, Wall PD, Nadvorna H, Steinbach T. Phantom limbs and related phenomena in recent traumatic amputations. Neurology. 1978 Mar;28(3):211-7. doi: 10.1212/wnl.28.3.211. PMID 564474
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777
- [Background] Hauschild M, Davoodi R, Loeb GE. A virtual reality environment for designing and fitting neural prosthetic limbs. IEEE Trans Neural Syst Rehabil Eng. 2007 Mar;15(1):9-15. doi: 10.1109/TNSRE.2007.891369. PMID 17436870
- [Background] Zeher MJ, Armiger RS, Burck JM, Moran C, Kiely JB, Weeks SR, Tsao JW, Pasquina PF, Davoodi R, Loeb G. Using a virtual integration environment in treating phantom limb pain. Stud Health Technol Inform. 2011;163:730-6. PMID 21335889